CLINICAL TRIAL: NCT00256698
Title: FACT: Anastrozole Monotherapy Versus Maximal Oestrogen Blockade With Anastrozole and Fulvestrant Combination Therapy; an Open Randomized, Comparative, Phase III Multicentre Study in Postmenopausal Women With Hormone Receptor Positive Breast Cancer in First Relapse After Primary Treatment of Localized Tumor.
Brief Title: Anastrozole Monotherapy Versus Maximal Oestrogen Blockade With Anastrozole and Fulvestrant Combination Therapy
Acronym: FACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6997L00002; 9238SW/0001; FACT
Record Dates: First submitted 2005-11-20; First posted 2005-11-22 (Estimated); Results first posted 2011-02-09 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: Hormone; receptor; positive; breast; cancer; first; relapse
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Recurrence | interventions — Fulvestrant; Anastrozole

ARMS (2):
- 1 (Active Comparator): Anastrozole
  Interventions: Drug: Anastrozole
- 2 (Experimental): Anastrozole + Fulvestrant
  Interventions: Drug: Fulvestrant; Drug: Anastrozole

INTERVENTIONS:
Drug: Fulvestrant — intramuscular injection 250 mg loading dose (LD) regimen
  Other Names: Faslodex; ZD9238
  Arms: 2
Drug: Anastrozole — 1 mg oral tablet
  Other Names: Arimidex; ZD1033

SUMMARY:
The purpose of this study is to determine the efficacy of anastrozole monotherapy versus maximal oestrogen blockade with combinated therapy of fulvestrant and anastrozole compared with in treatment of hormone receptor positive women with first relapse of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent, postmenopausal females, histological or cytological confirmed oestrogene and/or progesterone (PgR) receptor positive breast cancer, local recurrence or metastasis

Exclusion Criteria:

* Previous systemic endocrine therapy for advanced or recurrent disease; prior fulvestrant therapy
* Premenopausal women

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2004-01; Primary Completion 2009-04 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Henriksson, MD, Study Director — AstraZeneca
Locations (85):
- Canada (5):
  - Research Site, Brampton
  - Research Site, Halifax
  - Research Site, Kingston
  - Research Site, Ontario
  - Research Site, Toronto
- Research Site, San José, Costa Rica
- Finland (2):
  - Research Site, Hämeenlinna
  - Research Site, Turku
- France (9):
  - Research Site, Avignon
  - Research Site, Caen
  - Research Site, Créteil
  - Research Site, Grenoble
  - Research Site, La Chaussée-Saint-Victor
  - Research Site, Perpignan
  - Research Site, Périgueux
  - Research Site, Saint Cyr Sur Louire
  - Research Site, Toulouse
- Germany (24):
  - Research Site, Augsburg
  - Research Site, Cologne
  - Research Site, Düsseldorf
  - Research Site, Erlangen
  - Research Site, Frankfurt
  - Research Site, Gifhorn
  - Research Site, Großhadern
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Ingolstadt
  - Research Site, Kassel
  - Research Site, Kiel
  - Research Site, Leipzig
  - Research Site, Leverkusen
  - Research Site, Magdeburg
  - Research Site, Mannheim
  - Research Site, Marburg
  - Research Site, München
  - Research Site, Rostock
  - Research Site, Trier
  - Research Site, Ulm
  - Research Site, Ziwicken
- Research Site, Guatemala City, Guatemala
- Research Site, Reykjavik, Iceland
- Italy (9):
  - Research Site, Como
  - Research Site, Fabriano
  - Research Site, Ferrara
  - Research Site, Florence
  - Research Site, Lugo
  - Research Site, Milan
  - Research Site, Taormina
  - Research Site, Treviglio
  - Research Site, Vicenza
- Norway (7):
  - Research Site, Drammen
  - Research Site, Ilesund
  - Research Site, Oslo
  - Research Site, Porsgrunn
  - Research Site, Stavanger
  - Research Site, Troms
  - Research Site, Trondheim
- Portugal (4):
  - Research Site, Cascais
  - Research Site, Coimbra
  - Research Site, Lisbon
  - Research Site, Santa Maria da Feira
- Sweden (18):
  - Research Site, Halmstad
  - Research Site, Helsingborg
  - Research Site, Kalmar
  - Research Site, Karlskrona
  - Research Site, Kristianstad
  - Research Site, Link'ping
  - Research Site, M'lndal
  - Research Site, Malm
  - Research Site, Norrk'ping
  - Research Site, Skellefteå
  - Research Site, Skövde
  - Research Site, Södra Sunderbyn
  - Research Site, Stockholm
  - Research Site, Sundsvall
  - Research Site, Umeå
  - Research Site, V'rnamo
  - Research Site, V'stervik
  - Research Site, Varberg
- Turkey (Türkiye) (4):
  - Research Site, Ankara
  - Research Site, Edirne
  - Research Site, Gaziantep
  - Research Site, Istanbul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 258 patients were randomised to Fulvestrant + Anastrozole and 256 patients were randomised to Anastrozole. In each treatment group, there were 2 patients who did not receive any trial therapy and so have been excluded from the safety summaries.
Groups:
- Fulvestrant + Anastrozole: Fulvestrant 250 mg Loading Dose Regimen + Anastrozole 1 mg
- Anastrozole: Anastrozole 1 mg
Period: Overall Study
Arm/Group | Fulvestrant + Anastrozole | Anastrozole
Started | 258 | 256
Completed | 91 | 84
Not Completed | 167 | 172
Not completed — Withdrawal by Subject | 7 | 7
Not completed — Adverse Event | 13 | 6
Not completed — Protocol Violation | 6 | 5
Not completed — Lost to Follow-up | 1 | 3
Not completed — disease progression | 97 | 105
Not completed — still ongoing at data cut-off | 41 | 46
Not completed — withdrawn due to osteoporosis | 1 | 0
Not completed — Prematurely Discontinued | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fulvestrant + Anastrozole | Anastrozole | Total
Number analyzed (Participants) | 258 | 256 | 514
Age Continuous [Mean (Standard Deviation); unit: Years] | 65.2 (9.6) | 63.4 (10.3) | 64.3 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 258 | 256 | 514
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression (TTP)
Description: RECIST (Response Evaluation Criteria in Solid Tumours) assessments carried out every 8 weeks from randomisation until data cut-off on 30th April 2009. TTP, time in months to worsen 'progression' according to RECIST criteria. (RECIST is a set of published rules that define when cancer patients improve "respond", stay the same "stable"or worsen "progression" during treatments.
Time Frame: RECIST assessments carried out every 8 weeks from randomisation until data cut-off on 30th April 2009
Measure: Median (Full Range); unit: months
Arm/Group | Fulvestrant + Anastrozole | Anastrozole
Number analyzed (Participants) | 258 | 256
months | 10.8 [0 to 49.31] | 10.2 [0 to 54.34]

2. Secondary Outcome: Percentage of Evaluable Participants With Objective Response Rate (ORR)
Description: No. of patients who were objective responders over the no. of patients evaluable for response x100. An objective responder = a patient whose best response is either CR (disappearance of all lesions) or PR (>= 30% shrinkage in the sum of the longest diamemeters of the measurable lesions + no new lesions + no progression of non-measurable lesions)
Time Frame: RECIST tumour assessments carried out every 8 weeks from randomisation until data cut-off on 30th April 2009
Measure: Number; unit: Percentage of evaluable participants
Arm/Group | Fulvestrant + Anastrozole | Anastrozole
Number analyzed (Participants) | 129 | 113
Percentage of evaluable participants | 31.8 | 33.6

3. Secondary Outcome: Percentage of Clinical Benefit Rate (CBR) Responders
Description: No. of patients who were clinical benefit responders over the no. of randomised patients x100. A clinical benefit responder = a patient whose best response is CR, PR or SD>=24 weeks (where a best response of SD = no new lesions and for existing lesions; neither suffient shrinkage to count as PR nor sufficient growth to count as progression)
Time Frame: RECIST tumour assessments carried out every 8 weeks from randomisation until data cut-off on 30th April 2009
Measure: Number; unit: Percentage of participants
Arm/Group | Fulvestrant + Anastrozole | Anastrozole
Number analyzed (Participants) | 258 | 256
Percentage of participants | 55.0 | 55.1

4. Secondary Outcome: Duration of Response (DoR)
Description: Median time from randomisation until objective progression or death (in the absence of objective progression), measured only in those patients who are objective responders
Time Frame: RECIST tumour assessments carried out every 8 weeks from randomisation until data cut-off on 30th April 2009
Measure: Median (Full Range); unit: months
Arm/Group | Fulvestrant + Anastrozole | Anastrozole
Number analyzed (Participants) | 129 | 113
months | 22.3 [5.55 to 46.95] | 18.2 [7.20 to 49.77]

5. Secondary Outcome: Duration of Clinical Benefit (DoCB)
Description: Median time from randomisation until objective progression or death (in the absence of objective progression), measured only in those patients who are clinical benefit responders
Time Frame: RECIST tumour assessments carried out every 8 weeks from randomisation until data cut-off on 30th April 2009
Measure: Median (Full Range); unit: months
Arm/Group | Fulvestrant + Anastrozole | Anastrozole
Number analyzed (Participants) | 258 | 256
months | 18.5 [1.64 to 46.95] | 18.1 [5.19 to 54.34]

6. Secondary Outcome: Time to Treatment Failure (TTF)
Description: Time from randomisation until the date of discontinuation of randomised treatment for any reason
Time Frame: From randomisation until data cut-off on 30th April 2009
Measure: Median (Full Range); unit: months
Arm/Group | Fulvestrant + Anastrozole | Anastrozole
Number analyzed (Participants) | 258 | 256
months | 12.4 [0 to 46.95] | 11.4 [0 to 54.34]

7. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is equivalent to time to death. Time from randomisation until the date of death
Time Frame: All deaths occurring between randomisation and data cut-off on 30th April 2009 are included.
Measure: Median (Full Range); unit: months
Arm/Group | Fulvestrant + Anastrozole | Anastrozole
Number analyzed (Participants) | 258 | 256
months | 37.8 [0.07 to 61.86] | 38.2 [0.13 to 60.39]

ADVERSE EVENTS:
Arm/Group | Fulvestrant + Anastrozole | Anastrozole
Serious Adverse Events (participants affected / at risk) | 40/256 | 45/254
Other Adverse Events (participants affected / at risk) | 161/256 | 178/254
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fulvestrant + Anastrozole (N=256) | Anastrozole (N=254)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Cardiac Failure (Cardiac disorders) | 3 | 1
Pericardial Effusion (Cardiac disorders) | 0 | 2
Angina Pectoris (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial Flutter (Cardiac disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Ventricular Arrhythmia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
General Physical Health Deterioration (General disorders) | 0 | 3
Chest Pain (General disorders) | 1 | 2
Pain (General disorders) | 0 | 2
Fatigue (General disorders) | 2 | 1
Oedema Peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 2
Urinary Tract Infection (Infections and infestations) | 0 | 2
Infection (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 0 | 1
Viral Infection (Infections and infestations) | 0 | 1
Bronchpneumonia (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 2
Femur Fracture (Injury, poisoning and procedural complications) | 2 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 0
Fractured Sacrum (Injury, poisoning and procedural complications) | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 1 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 | 0
Blood Creatinine Increased (Injury, poisoning and procedural complications) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases To Meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 2
Syncope (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 1 | 1
Intracranial Haematoma (Nervous system disorders) | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 1
Cerebellar Infarction (Nervous system disorders) | 1 | 0
Cerebral Infarction (Nervous system disorders) | 1 | 0
Peripheral Motor Neuropathy (Nervous system disorders) | 1 | 0
Spinal Cord Compression (Nervous system disorders) | 1 | 0
Syncope Vasovagal (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Foot Amputation (General disorders) | 0 | 1
Venous Stasis (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fulvestrant + Anastrozole (N=256) | Anastrozole (N=254)
Nausea (Gastrointestinal disorders) | 23 | 27
Constipation (Gastrointestinal disorders) | 15 | 12
Diarrhoea (Gastrointestinal disorders) | 15 | 13
Vomiting (Gastrointestinal disorders) | 13 | 9
Fatigue (General disorders) | 27 | 33
Urinary tract infection (Infections and infestations) | 14 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 | 27
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 9
Hot flush (Vascular disorders) | 21 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that they cannot disclose or publish any information to do with the trial without consent from AstraZeneca